CLINICAL TRIAL: NCT05494255
Title: The Effects of Pre-extubation Single Recruitment Maneuver on Lung Ultrasound Scores and Postoperative Oxygenation in Laparoscopic Nephrectomy Surgeries
Brief Title: The Effects of Pre-extubation Single Recruitment Maneuver on Perioperative Atelectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emre Sertaç Bingül, Principal investigator, Lecturer, Medical Doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2022/1066
Record Dates: First submitted 2022-08-06; First posted 2022-08-09 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group RM (Active Comparator): One single recruitment maneuver will be applied in this group at the end of the surgery and before the extubation
  Interventions: Other: Recruitment maneuver
- Group NoRM (No Intervention): Usual care will be applied in this group

INTERVENTIONS:
Other: Recruitment maneuver — In Group RM (intervention group) after skin closure, mechanical ventilation settings will be set to FiO2:100%, I:E=1:1, respiratory rate: 6, and then tidal volume will be increased gradually by 150 ml until reaching a plato pressure of 30 mmHg. After 3 breaths in this state, RM will be considered accomplished. LUS evaluation will be made just before and after the RM.
  Arms: Group RM

SUMMARY:
Laparoscopic surgeries may cause atelectasis on the lungs which may stay clinically occult after the surgery. Lung Ultrasound Scoring (LUS) can provide an objective measuring system to understand the condition of the lungs in the perioperative period. In this randomized controlled study, it is aimed to investigate the effects of one single recruitment maneuver (RM) just before emergence and extubation (at the end of surgery) on LUS scores and postoperative recovery room oxygenation in laparoscopic nephrectomy surgeries. Accordingly, the intervention group will be applied single RM before extubation, while the control group will be awaken without RM.

There will be LUS evaluation at 4 different time for intervention group (Group RM) points that are:

T1: 5 min after the intubation T2: At the end of surgery (After skin closure, before recruitment maneuver) T3(RM): After recruitment maneuver, before extubation T4: 30 minutes after extubation in the recovery room

LUS evaluation will be made at 3 different time points in control group (Group NoRM):

T1: 5 min after the intubation T3(NoRM): Before extubation (no recruitment maneuvers will be made) T4: 30 minutes after extubation in the recovery room.

The primary outcome is the comparison of the T3 LUS scores. Assuming a 40% difference in the T3 LUS score, total number of 30 patients were calculated to be included in the study with an alpha value of 0.05 and 95% power. A possible drop-out of 5 patients per group, 20 patients were planned to be enrolled in each group.

Secondary outcomes will include; difference in T4 LUS scores, the effect of RM on postoperative recovery room oxygenation, and the effect of deltaLUS (T3-T2) on postoperative recovery room oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Laporoscopic nephrectomy patients who will be operated in lateral positions
* Elective, semi-elective surgeries

Exclusion Criteria:

* Patients with emphysema
* Patients with documanted heart failure
* Patients requiring intraoperative multiple recruitment maneuver due to hypoxemia
* Patients with hemodynamic instability
* Patients with pneumothorax risk
* Emergency surgery
* Patients requiring intraoperative liberal fluid therapy (>10 cc/kg/hr)
* Patients requiring blood products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Comparison of the pre-extubation LUS scores (T3) | Up to 4 hours
  Lung ultrasound will be applied in each group to observe the lungs' condition (atelectasis,consolidation...) and understand the effect of a "single" recruitment maneuver. To obtain LUS score; each lobe is examined on 6 different areas which will be scored from 0 to 3, and both lungs will be evaluated. Therefore maximum score may change from 0 (no atelectasis, best condition) to 36 (worst condition, broad atelectasis and consolidation).

SECONDARY OUTCOMES:
Comparison of recovery room LUS scores (T4) | Up to 4.5 hours
  Lung ultrasound will be applied at post-extubation 30th minute to evaluate the compare the groups for the possible effect of single RM. To obtain LUS score; each lobe is examined on 6 different areas which are scored from 0 to 3, and both lungs will be evaluated. Therefore maximum score may change from 0 (no atelectasis, best condition) to 36 (worst condition, broad atelectasis and consolidation).
Comparison of recovery room PaO2 | Up to 4.5 hours
  Arterial blood gas will be analyzed at post-extubation 30th minute along with LUS to observe the effect of RM on oxygenation
The effect of deltaLUS (T3-T2) on oxygenation | Up to 4.5 hours
  DeltaLUS values will be analyzed for relation with post-extubation 30th min PaO2 values.
Length of stay in post anesthesia care unit (PACU) | Up to 4 hours
  The duration required for the patient to stay in PACU (minutes)
Length of stay in hospital | Up to 2 weeks
  The duration required for patient to stay in hospital (days)
Postoperative respiratory complications | Up to 5 days
  Incidence of mild-to-severe respiratory failure, pneumothorax, ALI, ARDS, bronchospasm, pneumonia
Predictive value of dependant lung T3 (preextubation) LUS score detecting postoperative pulmonary complications | Up to 24 hours
  Sensitivity and specifity (Area under the curve-ROC analysis) values of LUS score of dependant lung. (0=the best condition of the dependant lung, 18=the worst condition of the dependant lung with consolidation and atelectasis)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request